CLINICAL TRIAL: NCT01552473
Title: Brain Training to Enhance Frontal Lobe Reasoning in Soldiers and Civilian Adults With TBI
Brief Title: Brain Training to Enhance Frontal Lobe Reasoning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Dallas (Other)
Collaborators: University of Texas Southwestern Medical Center (Other); Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dan Krawczyk, Professor, The University of Texas at Dallas
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU 032011-191
Record Dates: First submitted 2012-03-06; First posted 2012-03-13 (Estimated); Results first posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Traumatic Brain Injury
Keywords: TBI; Traumatic Brain Injury; combat related injury; blast injury; concussion; sleep problems; attention problems; memory problems; headaches; dizziness; OEF; OIF; Veterans; Civilian
MeSH Terms: conditions — Brain Injuries, Traumatic; Blast Injuries; Brain Concussion; Parasomnias; Memory Disorders; Headache; Dizziness

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Brain Training Program 1 (Active Comparator): Training Program focusing on providing educational information of cognitive issues related to TBI
  Interventions: Behavioral: Brain Training Program 1
- Brain Training Program 2 (Experimental): Program focuses on strategies to address cognitive issues following TBI
  Interventions: Behavioral: Brain Training Program 2

INTERVENTIONS:
Behavioral: Brain Training Program 1 — The training program includes 12 sessions conducted over 8 weeks. The goal of these treatment sessions is to provide information on brain injury and its recovery process. Activities involved in the sessions include discussion of study material. Participants will be encouraged to apply the information to their daily lives. The program includes additional outside practice of the activities.
  Arms: Brain Training Program 1
Behavioral: Brain Training Program 2 — The training program includes 12 sessions conducted over 8 weeks. The goal of these treatment sessions is to provide strategies to improve brain injury and its recovery process. Activities involved in the sessions include strategies and discussion of study material. Participants will be encouraged to apply the strategies and information to their daily lives. The program includes additional outside practice of the activities.
  Arms: Brain Training Program 2

SUMMARY:
This study is being done to improve the ability to diagnose and to achieve higher-levels of functional recovery in soldiers and civilians who have suffered either mild Traumatic Brain Injury (TBIs) or moderate-to-severe TBIs at chronic stages of brain recovery (greater than 12 months).

DETAILED DESCRIPTION:
In the current randomized control trial, we study the efficacy of a functionally relevant cognitive training program applied to individuals who are experiencing the effects of chronic TBI. The top-down training program labeled SMART (Strategic Memory Advanced Reasoning Training) adopts an integrative approach to train functionally relevant complex reasoning abilities (versus specific skills). This integrative approach focused on frontal lobe functions has shown promising results in a preliminary study. SMART is compared to an equally engaging education-based program labeled BHW (Brain Health Workshop). Both SMART and BHW are short-term, intensive (18 h of training over 8 weeks) group training programs that are comparable with regard to training time, amount of information, group discussions, and homework assignments. The overall goal of this trial is to examine how training integrative frontal lobe-mediated processes might improve functioning in brain injury survivors, including military service and civilian populations. We include a range of individuals with different injury types and functional abilities. We use a broad variety of assessment tools, including cognitive, neuroimaging, and functional measures, to compare the training groups.

Our overall goal is to improve the fidelity of TBI diagnoses and to achieve higher levels of functional recovery in soldiers and civilians who have suffered mild to moderate TBIs and are at the chronic stage of brain recovery. This study is also to determine the efficacy of an empirically and theoretically driven framework to enhance frontal lobe-mediated reasoning ability in individuals with TBI, given a relatively short training duration, on trained and untrained cognitive skills, on brain changes, and on measures of real-life function. Toward these aims, this trial is enrolling both soldiers and civilians with a TBI (approximately 50 mild and 50 moderate chronic TBI patients). We use cognitive tests (assessing memory, reasoning, and comprehension abilities), functional MRI scans (performing tests of cognitive function while the subject is receiving an MRI scan), and white matter maps constructed using diffusion tensor imaging (DTI) scans. The MRI scans will be used to provide biomarkers of the contributions of different brain regions to performing cognitive tasks (e.g., memory, reasoning, etc.), as well as assessments of brain efficiency, functional brain connectivity, and brain morphology. We use these measurements to gain an understanding of each individual's cognitive skills and neural measures prior to cognitive intervention. These measures also serve as indicators of the baseline function of each soldier or civilian, to be compared with after intervention, at which point they undergo post-training cognitive, MRI, and DTI assessments, enabling us to make outcome comparisons between the two different cognitive interventions. Finally, we conduct a follow-up assessment with neuropsychological and cognitive measures and neuroimaging 3 months after the interventions to assess how individuals maintain any functional changes that may occur because of the cognitive interventions.

We are targeting this intervention toward mild and moderate TBI participants, who have relatively high functioning skills. The demands of the training can be too high for some individuals falling into the more severe range, in the frequency, duration, and type of strategies and skills emphasized. We also aim to address the high level of need placed upon studies of milder TBI cases, particularly with military populations. This priority is also emphasized by the sponsoring agency, the US Department of Defense, advocating for more studies of mild TBI under the funding mechanism supporting this work.

ELIGIBILITY:
Inclusion Criteria:

* 19-65 years of age
* Sustained a traumatic brain injury at least 6 months previously
* Comprehend simple instructions, perform tasks and take part in intervention
* Read, speak and comprehend English
* Participate in tasks involving motor abilities such as use of at least one arm or hand

Exclusion Criteria:

* Not proficient in reading, comprehending or speaking English
* Pre-existing Cerebral Palsy, Mental Retardation, Autism, Epilepsy, Schizophrenia, or Pervasive Developmental Disorder
* Individuals with Psychosis, Active Behavioral Disorder, or uncontrolled epilepsy
* Women who are pregnant

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2012-03; Primary Completion 2015-07 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Krawcyzk, Ph.D., Principal Investigator — University of Texas
Locations (1):
- Center for BrainHealth, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Krawczyk DC, Marquez de la Plata C, Schauer GF, Vas AK, Keebler M, Tuthill S, Gardner C, Jantz T, Yu W, Chapman SB. Evaluating the effectiveness of reasoning training in military and civilian chronic traumatic brain injury patients: study protocol. Trials. 2013 Jan 30;14:29. doi: 10.1186/1745-6215-14-29. PMID 23363480
- See also: Center for BrainHealth — http://centerforbrainhealth.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Brain Health Workshop (BHW): A comparison-training program in cognitive training trials. The topics are presented with information (via Power Point) relevant to the participants' health and brain injury. Specifically, anatomy, functioning of each lobe of the brain, neurotransmitters, effects of TBI on cognitive functioning, and general principles of neuroplasticity. Other sessions pertain to the effects of sleep, diet, exercise, and social bonds on the brain.
- Strategic Memory Advanced Reasoning Training (SMART): The SMART protocol trains a common set of three multidimensional and inter-related strategies to apply to a wide range of everyday tasks. The strategies draw upon top-down processes to improve cognitive control functions, including strategic attention, integrative reasoning and innovation.
  Strategic attention strategies focus on intentional management of input by blocking distractions and irrelevant input, and factoring in regular mental breaks. The negative toll of multitasking on cognitive performance and productivity is integral to strategic attention. Integrative reasoning strategies build on strategic attention to engage in synthesis, abstraction, and implementation processes. Abstracting meanings (or ideas) from input/data to understand big ideas, take-home messages, and meaningful goals (that can be implemented) forms the core of this second part of the training.
Period: Pre-training Testing
Arm/Group | Brain Health Workshop (BHW) | Strategic Memory Advanced Reasoning Training (SMART)
Started | 52 | 56
Completed | 52 | 56
Not Completed | 0 | 0
Period: Post-training Testing
Arm/Group | Brain Health Workshop (BHW) | Strategic Memory Advanced Reasoning Training (SMART)
Started | 52 | 56
Completed | 35 | 38
Not Completed | 17 | 18
Period: Delayed Post-training Testing
Arm/Group | Brain Health Workshop (BHW) | Strategic Memory Advanced Reasoning Training (SMART)
Started | 35 | 38
Completed | 35 | 35
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Brain Health Workshop (BHW): The BHW program focuses on teaching facts about brain functions and influences on cognition. This program was originally developed at the Rotman Institute, Canada [34]. The BHW includes topics such as an overview of brain anatomy, neuroplasticity, memory, attention and executive functions, aging and the brain, sleep and stress, diet and physical exercise, and social bonds and the brain. We adapted the curriculum to approximate the general structure of SMART training, including matching for the number of sessions, duration, discussions, and homework assignments.
- Strategic Memory Advanced Reasoning Training (SMART): SMART utilizes a strategy-based approach to train individuals in abstract thinking ability. Specifically, participants are trained in cognitive control strategies of strategic attention, integration, and innovation, which facilitate abstraction abilities. Strategic attention involves blocking less relevant details to focus on important information. Integration incorporates strategies to abstract and create meanings or goals from information or tasks. Innovation focuses on generating and discovering novel concepts, ideas, and diverse goals and perspectives. The strategy instruction is hierarchical, with each strategy dynamically building upon previous strategies. The SMART program incorporates a wide range of discourse and task materials relevant in daily life contexts, such as planning an event, going on a job interview, learning from a lecture, or explaining a concept.
- Total: Total of all reporting groups
Arm/Group | Brain Health Workshop (BHW) | Strategic Memory Advanced Reasoning Training (SMART) | Total
Number analyzed (Participants) | 52 | 56 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.19 (13.37) | 40.59 (13.05) | 41.36 (13.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 41
  Male | 32 | 35 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 45 | 51 | 96
  Unknown or Not Reported | 4 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 8 | 14
  White | 42 | 47 | 89
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 0 | 4
Years of Education [Mean (Standard Deviation); unit: years] | 16.34 (3.07) | 15.80 (2.43) | 16.05 (2.74)
Socio-economic Status (SES) [Mean (Standard Deviation); unit: units on a scale] — This measures social class, especially social class of origin identity. The score range is 8 (lowest socioeconomic status) to 66 (highest socioeconomic status) in weighted units indicating categories of economic achievement from one's lifespan. This score is ordinal only and does not intend to describe or define an individual's social or economic standing in the community. It is sufficient for regression analysis or for creating social status groups based on the data collected.
  units on a scale | 44.81 (13.09) | 40.44 (14.85) | 42.48 (14.16)
Civilian/Military [Count of Participants; unit: Participants]
  Civilian | 21 | 31 | 52
  Military (Veteran) | 31 | 25 | 56
Marital Status [Count of Participants; unit: Participants]
  Married | 22 | 17 | 39
  Single | 23 | 29 | 52
  Widow | 1 | 0 | 1
  Divorced | 4 | 10 | 14
  Separated | 2 | 0 | 2
Current IQ [Mean (Standard Deviation); unit: units on a scale] | 109.94 (12.42) | 107.93 (10.23) | 108.84 (11.25)
Type of Head Injury [Count of Participants; unit: Participants]
  Blast | 6 | 6 | 12
  Blunt-force trauma | 9 | 5 | 14
  Falls | 6 | 9 | 15
  Multiple Injuries | 7 | 11 | 18
  Sports | 4 | 11 | 15
  Vehicular Accident(s) | 16 | 14 | 30
  Unknown | 4 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Glasgow Outcome Scale-Extended
Description: Assesses disability after brain injury (1 dead to 8 good recovery). A higher score is a better outcome.
Time Frame: Pre-training (Baseline) Neuropsychological Test
Population: Community dwelling individuals between the ages of 19 and 65 years with a history of chronic TBI (> 6 months post-injury).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Brain Health Workshop (BHW) | Strategic Memory Advanced Reasoning Training (SMART)
Number analyzed (Participants) | 52 | 56
units on a scale | 6.21 (0.75) | 6.30 (0.76)

2. Primary Outcome: Community Integration Questionnaire
Description: To examine short-term effects of treatment on cognition and real-life outcomes relating to how successful someone is able to integrate within their community (0 lowest integration (worst outcome) to 40 maximal integration (best outcome)). A higher score is a better outcome.
Time Frame: Neuropsychological changes from baseline to 10 weeks post-training
Population: Community dwelling individuals (41 women and 67 men) between the ages of 19 and 65 years with a history of chronic TBI (> 6 months post-injury).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Brain Health Workshop (BHW) | Strategic Memory Advanced Reasoning Training (SMART)
Number analyzed (Participants) | 47 | 56
units on a scale | 16.91 (5.04) | 18.71 (5.08)

3. Primary Outcome: Functional Status Exam
Description: To examine short-term effects of treatment on outcomes. - (0 highest function (best outcome) to 31 lowest function (worst outcome)). A lower score is a better outcome.
Time Frame: Measure at 10 weeks post-training
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Brain Health Workshop (BHW) | Strategic Memory Advanced Reasoning Training (SMART)
Number analyzed (Participants) | 48 | 56
units on a scale | 24.02 (6.93) | 22.14 (6.23)

4. Primary Outcome: Daneman-Carpenter Reading Span Test
Description: Scored as 0 words to 7 words comprehended. Higher scores indicate better comprehension and thus a better outcome. Lower scores indicates a lower degree of comprehension. A higher score is a better outcome.
Time Frame: Measure at 10 weeks post-training
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Brain Health Workshop (BHW) | Strategic Memory Advanced Reasoning Training (SMART)
Number analyzed (Participants) | 48 | 55
units on a scale | 2.81 (0.89) | 2.89 (1.07)

5. Primary Outcome: Hayling Sentence Completion Test
Description: To examine short-term effects of treatment on cognition by working memory. The Hayling Sentence Completion test measures response initiation (range 0 best to 30 worst). A lower score is a better outcome.
Time Frame: Measure at 10 weeks post-training
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Brain Health Workshop (BHW) | Strategic Memory Advanced Reasoning Training (SMART)
Number analyzed (Participants) | 48 | 56
units on a scale | 5.96 (1.22) | 6.05 (1.35)

6. Primary Outcome: Awareness Questionnaire
Description: To examine short-term effects of treatment on real-life outcomes. This test measures impaired self-awareness after brain injury. The scale ranges from 17 (lowest self-awareness level, worst outcome) to 85 (highest self-awareness level, best outcome). A higher score is a better outcome.
Time Frame: Measure at 10 weeks post-training
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Brain Health Workshop (BHW) | Strategic Memory Advanced Reasoning Training (SMART)
Number analyzed (Participants) | 48 | 56
units on a scale | 34.94 (9.08) | 38.00 (9.48)

7. Secondary Outcome: Network Based Statistics in Brain Connectivity
Description: Brain network connectivity from functional brain imaging was computed using Network-Based Statistics. Data were adjusted to form one number to characterize the significant connection changes associated with the training. This was accomplished by computing a change score. This change score combined the post-training (10 weeks), and 3-months post-training imaging data and compared that to the baseline (pre-training imaging data). This measure allows for an estimation of the number of statistically increased connections observed between different areas of the brain. A higher score indicates more significant connections and is considered to be a better outcome.
Time Frame: MRI measures taken at 10 weeks and 3 months post-training are combined and compared to baseline MRI yielding one number
Population: The participants included in this analysis completed Magnetic Resonance Imaging Scans. This analysis does not include all 108 participants. Some participants data were not included due to the fact that they were not adequate for the analysis due to motion artifacts which severely affect this type of imaging measurement.
Measure: Number; unit: number of significant brain connections
Arm/Group | Brain Health Workshop (BHW) | Strategic Memory Advanced Reasoning Training (SMART)
Number analyzed (Participants) | 29 | 31
number of significant brain connections | 0 | 14
Statistical Analysis 1: Comparison: Brain Health Workshop (BHW) vs Strategic Memory Advanced Reasoning Training (SMART); A network-based statistics analysis was carried out to determine brain connectivity differences observed at time points two (initial post-intervention testing phase) and three (the final post-intervention phase) occurring three months post-intervention; Test type: Other — This is a functional Magnetic Resonance Imaging analysis. We aimed to determine whether functional brain network connectivity was equivalent between the two intervention arms prior to the interventions beginning. This was computed in significant numbers of connections between the two groups; p = 0.01, Network Based Statistics analysis — This is a p-value that is used in Network Based Statistics analysis for resting-state functional brain network data; This is a type of statistical analysis used to test for group differences among functional connectivity levels between two or more groups; pNBS = .0001 — This analysis evaluated monotonic changes from time point 1 (pre-intervention) to time points 2 (immediate post-intervention) and 3 (12 weeks post-intervention) that may have occurred between the SMART and BHW groups

8. Secondary Outcome: Beck Depression Inventory (BDI)
Description: To examine short-term effects of treatment on measures current depressive symptoms from 0 (no depressive symptoms (best outcome)) to 63 (maximum depressive symptoms (worst outcome)). A lower score is a better outcome.
Time Frame: Measure taken at 10 weeks post-training
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Brain Health Workshop (BHW) | Strategic Memory Advanced Reasoning Training (SMART)
Number analyzed (Participants) | 46 | 56
scores on a scale | 18.28 (12.51) | 18.41 (10.59)

9. Secondary Outcome: Post Traumatic Stress Disorder (PTSD) Checklist
Description: To examine short-term effects of treatment on self-reported measure of symptoms of posttraumatic stress disorder. The test ranges from 0 minimal stress symptoms to 80 maximum stress symptoms. A lower score is a better outcome.
Time Frame: Measure taken at 10 weeks post-training
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Brain Health Workshop (BHW) | Strategic Memory Advanced Reasoning Training (SMART)
Number analyzed (Participants) | 47 | 54
scores on a scale | 46.76 (18.03) | 44.09 (15.84)

10. Secondary Outcome: Alcohol, Smoking and Substance Involvement Screening Test
Description: To examine short-term effects of treatment on problem substance use. The range is from 0 low levels of problem substance use to 414 (maximum level of problem substance use). A lower score is a better outcome.
Time Frame: Measure taken at 10 weeks post-training
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Brain Health Workshop (BHW) | Strategic Memory Advanced Reasoning Training (SMART)
Number analyzed (Participants) | 47 | 56
scores on a scale | 19.40 (15.50) | 22.18 (19.12)

11. Secondary Outcome: Alcohol Use Disorders Identification Test
Description: To examine short-term effects of treatment on real-life outcomes on alcohol use disorder. The test ranges from 0 lowest use (best outcome) to 40 maximal use (worst outcome). A lower score is a better outcome.
Time Frame: Measure taken at 10 weeks post-training
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Brain Health Workshop (BHW) | Strategic Memory Advanced Reasoning Training (SMART)
Number analyzed (Participants) | 47 | 56
scores on a scale | 2.94 (3.78) | 3.39 (4.12)

12. Secondary Outcome: Digit Vigilence Test
Description: To examine short-term effects of treatment on attention. The test is scored as time in seconds with the lowest amount of time indicating the best performance. A lower score is a better outcome.
Time Frame: Measure taken at 10 weeks post-training
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Brain Health Workshop (BHW) | Strategic Memory Advanced Reasoning Training (SMART)
Number analyzed (Participants) | 47 | 56
seconds | 413.06 (99.06) | 359.20 (72.74)

13. Secondary Outcome: Connor-Davidson Resilience Scale
Description: To examine short-term effects of treatment on resilience. the scores range from 0 (lowest reslience and worst outcome) to 100 (highest resilience and best outcome). A higher score is a better outcome.
Time Frame: Measure taken at 10 weeks post-training
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Brain Health Workshop (BHW) | Strategic Memory Advanced Reasoning Training (SMART)
Number analyzed (Participants) | 47 | 56
scores on a scale | 61.26 (12.86) | 64.38 (22.40)

14. Secondary Outcome: Wechsler Memory Scale
Description: To examine short-term effects of treatment on memory. The scores range from 0 (lowest memory level) to 20 (higher memory level). A higher score is a better outcome.
Time Frame: Measure taken at 10 weeks post-training
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Brain Health Workshop (BHW) | Strategic Memory Advanced Reasoning Training (SMART)
Number analyzed (Participants) | 48 | 56
scores on a scale | 12.96 (4.05) | 12.79 (4.08)

15. Secondary Outcome: Wechsler Abbreviated Scale of Intelligence Vocabulary Scale
Description: To examine short-term effects of treatment on vocabulary ability Score ranges from 20 (a lower level of vocabulary) to 80 (a higher level of vocabulary). A higher score is a better outcome.
Time Frame: Measure taken at 10 weeks post-training
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Brain Health Workshop (BHW) | Strategic Memory Advanced Reasoning Training (SMART)
Number analyzed (Participants) | 48 | 56
scores on a scale | 61.44 (7.84) | 58.14 (8.14)

16. Secondary Outcome: Wechsler Abbreviated Scale of Intelligence Matrix Reasoning
Description: To examine short-term effects of treatment on cognition with fluid reasoning being the measure ranging from 20 (lowest performance) to 80 (highest performance). A higher score is a better outcome.
Time Frame: Measure taken at 10 weeks post-training
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Brain Health Workshop (BHW) | Strategic Memory Advanced Reasoning Training (SMART)
Number analyzed (Participants) | 48 | 56
scores on a scale | 26.56 (4.30) | 27.64 (4.68)

17. Secondary Outcome: Wechsler Abbreviated Scale of Intelligence Similarities
Description: To examine short-term effects of treatment on cognition with a score of 20 indicating lowest similarities performance to 80 indicating the highest similarities performance. A higher score is a better outcome.
Time Frame: Measure taken at 10 weeks post-training
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Brain Health Workshop (BHW) | Strategic Memory Advanced Reasoning Training (SMART)
Number analyzed (Participants) | 48 | 56
scores on a scale | 37.69 (4.39) | 36.96 (3.71)

18. Secondary Outcome: Satisfaction With Life Scale
Description: To examine short-term effects of treatment on real-life outcomes. This ranges from 5 lowest satisfaction with life to 35 highest satisfaction with one's life. A higher score is a better outcome.
Time Frame: Measure taken at 10 weeks post-training
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Brain Health Workshop (BHW) | Strategic Memory Advanced Reasoning Training (SMART)
Number analyzed (Participants) | 48 | 56
scores on a scale | 17.56 (7.60) | 16.54 (7.85)

ADVERSE EVENTS:
Time Frame: Each participant was involved in the study for a total of twenty-one weeks. This consisted of one week during which the first assessment took place followed by eight weeks of cognitive intervention training in either of the two arms of the study and the first post-training assessment). Lastly, there was one additional testing session carried out twelve weeks after the completion of the training (and the first post-training assessment).
Description: No participants experienced adverse events, or serious adverse events.
Groups:
- Strategic Memory Advanced Reasoning Training Group: A group that experienced a cognitive intervention aimed at improving attention, memory, and reasoning skills.
- Brain Health Workshop: A group that experienced a cognitive intervention aimed at informing people about facts regarding the brain.
Arm/Group | Strategic Memory Advanced Reasoning Training Group | Brain Health Workshop
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/52
Other Adverse Events (participants affected / at risk) | 0/56 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes